CLINICAL TRIAL: NCT01072942
Title: Randomized, Single-blinded, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pulmonary Deposition, Pharmacokinetics and Pharmacodynamics of Ciprofloxacin in Japanese Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD; GOLD II-III), Following Multiple Inhalation of Ciprofloxacin PulmoSphere Inhalation Powder
Brief Title: To Evaluate the Safety, Tolerability, Pulmonary Deposition, Pharmacokinetics and Pharmacodynamics of Ciprofloxacin Inhale in Japanese Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD, GOLD II-III)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14019
Record Dates: First submitted 2010-01-27; First posted 2010-02-22 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive; Phase I; Pharmacokinetics; Microbiology
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Ciprofloxacin (Cipro InhaIe, BAYQ3939)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciprofloxacin (Cipro InhaIe, BAYQ3939) — Ciprofloxacin Inhale 50 and 75 mg 2 times a day (BID) for 10 days
  Arms: Arm 1
Drug: Placebo — Placebo TID for 10 days
  Arms: Arm 2

SUMMARY:
The study will be conducted in a single-center, randomized, single-blinded, placebo-controlled, dose escalation design with two dose groups.Multiple-dose inhalation of Ciprofloxacin inhale 50 and 75 mg or placebo will be administered to 16 Japanese patients with COPD in totalPatients with moderate to severe COPD, stage II or III according to GOLD criteria, will participate in the study.The study will consist of 2 steps as indicated below; starting at Step 1 (50 mg) and escalating doses up to Step 2 (75 mg), after the tolerability of the dose in the previous step is confirmed. In each step, the study will be conducted as multiple dose study with b.i.d. regimen for 10 days (between day 2 and 11) in a randomized, single-blind, placebo-controlled design. In addition, before and after the multiple dose administration, single administration will be conducted in each subject (day 0 and 12).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with COPD, 40 to 80 years of age
* All patients must have a diagnosis of COPD and must meet the following spirometric criteria: Patients must have relatively stable airway obstruction with a post-bronchodilator 30% </= Forced Expiratory Volume (FEV1) </= 65% of predicted normal. And a post-bronchodilator FEV1 / Forced Vital Capacity (FVC) <70%.

Exclusion Criteria:

* Patients with a significant respiratory disease other than COPD. A significant disease is defined as a disease which, in the opinion of the investigator
* Patients with a medical disorder, condition or history of such that would impair the patients ability to participate or complete this study in the opinion of the investigator, patients who have mental disorder which is inappropriate to communal living in a participation in a clinical study, who have no ability to give informed consent, or who have physical disability
* Patients with a history of CF
* Patients with clinically evident bronchiectasis
* Patients with a history of asthma
* Patients who have undergone thoracotomy with pulmonary resection
* Patients with relevant conspicuous findings in medical history and pre-study examination not related to the underlying disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Adverse event collection | Up to 3 weeks

SECONDARY OUTCOMES:
Microbiological examination | 14 days
Ciprofloxacin concentration in sputum | 14 days
Ciprofloxacin concentration in plasma | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Yufu, Oita Prefecture, Japan